CLINICAL TRIAL: NCT04235400
Title: Multimodal Analysis of Ocular Surface for Screening Dry Eye Disease
Brief Title: Multimodal Screening of Dry Eye Disease
Acronym: MAOS-S
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP191122; 2019-A03086-51 (Other: ID-RCB)
Record Dates: First submitted 2020-01-17; First posted 2020-01-21 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Dry Eye Disease
Keywords: dry eye; TBUT; NIBUT
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient with dry eye disease
  Interventions: Diagnostic Test: No Dye BreakUp Time

INTERVENTIONS:
Diagnostic Test: No Dye BreakUp Time — Measurement without dye of the tear meniscus height (TMH) which give an rapid hint on the quantity of tears present on the ocular surface, the measure in real time of the tear osmolarity and, at last, the analysis of the thickness of the tear's layer by interferometry (measurement of the light fringes reflected by the tears when illuminated with polarized light, whereby the complete layer or the lipid layer alone can be evaluated separately depending on the machines used) and of the assessment of the quality of the Meibomian glands (non-contact imaging by infrared illumination).

SUMMARY:
Two methods allow to evaluate tear breakup time (BUT): without prior dye instillation (No Dye BreakUp Time NDBUT) or after fluorescein instilation (FBUT). The interconnections between those two values are unknown

DETAILED DESCRIPTION:
To date, there are a limited numbers of tests available for screening ocular dryness:

i) assessement of tear production through Schirmer's test (paper strips are inserted into the eye for 5 minutes to measure the production of tears: normal value is superior to 15 mm wetting of the paper after 5 minutes, pathologic if inferior to 5-10 mm) ii) assessment of the ocular surface damage after instillation of fluorescein (presence of punctuate superficial lesions on the corneal and conjunctival epithelium) the with the slit lamp + blue filter iii) assessment of the FBUT (measurement of the tear breakup time after fluorescein dye instillation): normal value is superior to 15 seconds, pathologic value inf inferior to 5-10 seconds iv) assessment of the inflammation of eyelids (with the slit lamp). These diagnostic tests are used in everyday clinical practice, but however the international consensus conference (Dry Eye Workshop II, 2017) clearly recommended that, whenever practicable, some other tests must be carried out to optimize the efficacy the diagnostic procedure of dry eye disease. This is the case for the NDBUT (in opposition to the FBUT which uses fluorescein), the tear meniscus height (TMH) which give an rapid hint on the quantity of tears present on the ocular surface, the measure in real time of the tear osmolarity and, at last, the analysis of the thickness of the tear's layer by interferometry (measurement of the light fringes reflected by the tears when illuminated with polarized light, whereby the complete layer or the lipid layer alone can be evaluated separately depending on the machines used) and of the assessment of the quality of the Meibomian glands (non-contact imaging by infrared illumination).

All these techniques are recommended for the detection and the analysis of the mechanism inducing ocular dryness because they are non-invasive and painless. They also are recommended to be carried out jointly because there is still no single objective criterion that is sufficiently robust to be used alone to make this diagnosis, which is therefore ultimately based on an overall analysis of these various parameters.

Furthermore, the nature of the relationships between these different objective diagnostic tests remains still poorly understood.

One of the least well elucidated points in this respect is the relationship between the FBUT and the NDBUT, the latter having the theoretical advantage of being less subjective (the measurement is made by a medical device that detects the deformation time of a light test pattern projected onto the tear film). This method therefore tends to measure rather the moment when the film becomes thinner (generating the deformation of the test pattern), whereas the measurement of FBUT (i.e. after instillation of fluorescein), is certainly subjective but it measures the real tear break time, which corresponds physiologically to a critical moment (regulated by the blink reflex when sensitivity is normal). A retrospective study, carried out in patients known to suffer from dry eye disease and using many of the same instruments as those to be used in the present study, suggested that the NDBUT is generally longer than the FBUT (with an increasing difference with the values), which could be considered paradoxical (the thinning being expected to precede the complete rupture). This relationship must therefore be studied prospectively to analyze the nature of this difference (correlation?) and its relationship with other markers of dry eye disease.

The level of subjective symptoms and the impact on the quality of life felt by the patient will be recorded in order to explore whether the possible difference between NDBUT and FBUT is correlated with the intensity and/or frequency of the symptoms felt.

ELIGIBILITY:
Inclusion Criteria:

* adult patient (age >18 yo),
* known allergy to topical fluorescein
* Patient informed of the study who gave it's non-opposition to participate

Exclusion Criteria:

* Ocular surgery (including punctal plugs surgery) within the 3 previous months
* contact lens wearing within the 3 previous months
* Patient under guardianship or convicted person
* pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major patients consulting for dry eyes or requiring dry eye screening
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-01-28 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
results of the NDBUT and FBUT | at the end of the study (1year)
  analysis of the interconnections between the measure of the tear breakup time without adjunction of dye and measure obtained after instillation of the dye (fluorescein)

SECONDARY OUTCOMES:
Ocular Surface Disease Index (OSDI) questionnaire results | at day 1
  to assess the symptoms of ocular dryness
visual analogic scale (EVA) for the assessment of the impact of the dry eye for the patient | at day 1
  0 means no impact, 100 means total impact of the disease
Tear meniscus height | at day 1
  with the LACRYDIAG device
Results of the tears interferometry with the LACRYDIAG device | at day 1
Results of the tears interferometry with the LIPIVIEW device | at day 1
Results of the meibography with the LIPIVIEW device | at day 1
Thickness of the lipidic layer measured with LIPIVIEW device | at day 1
Tear osmolarity | at day 1
  normal osmolarity is about 290 milliosmol per liter (mOsm/l). An elevated reading, >313 mOsm/L indicates hyperosmolarity, and thus the loss of homeostasis leading to dry eye disease
Quality of the corneal epithelium (after fluorescein instillation, Oxford scale) | at day 1
Tear's production measured by Schirmer I test | at day 1
  normal value is superior to 15 mm wetting of the paper after 5 minutes, pathologic if inferior to 5-10 mm

CONTACTS AND LOCATIONS:
Overall Officials: Marc LABETOULLE, Pr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Opthtalmology Departement, Bicêtre Hospital, Le Kremlin-Bicêtre, Val De Marne, France

IPD SHARING:
Plan to Share IPD: No